CLINICAL TRIAL: NCT02853136
Title: Influence of Fluvoxamine on the Pharmacokinetics of BI 409306 After Oral Administration (Randomized, Open-label, Two-treatment, Two-sequence, Two-period Crossover Study)
Brief Title: Influence of Fluvoxamine on the Pharmacokinetics of BI 409306
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1289.35; 2016-000752-10 (EudraCT Number)
Record Dates: First submitted 2016-07-29; First posted 2016-08-02 (Estimated); Results first posted 2024-08-21 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-03

CONDITIONS: Healthy
MeSH Terms: interventions — Fluvoxamine; Solutions; BI 409306

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- 3 mg BI 409306 [R1]/3 mg BI 409306 + 100 mg Fluvoxamine [T1] (Experimental): The subjects were administered 3 milligram [mg] BI 409306 Powder for Oral Solution [PfOS] single dose for one day in the pilot phase, taken as 6 mL of 0.5 mg/mL BI 409306 solved in 5 mg/mL [milliLiter] tartaric acid orally with 240 mL of water after an overnight fast of at least 10h, followed by 3 mg BI 409306 PfOS single dose for one day together with 100 mg Fluvoxamine [Fevarin®] film-coated tablet once daily orally with 240 mL of water after an overnight fast of at least 10h.
  Prior to the combined treatment, Fluvoxamine was given for 3 days: 50 mg twice daily on Day -3, followed by 100 mg bid on Day -2 and Day -1.
  There was a washout of at least 3 days after administration of BI 409306 in R1.
  Interventions: Drug: Fluvoxamine; Drug: BI 409306 - Powder for oral solution (PfOS)
- 3 mg BI 409306 + 100 mg Fluvoxamine [T1]/3 mg BI 409306 [R1] (Experimental): The subjects were administered 3 mg BI 409306 PfOS single dose for one day in the pilot phase together with 100 mg Fluvoxamine [Fevarin®] film-coated tablet once daily orally with 240 mL of water after an overnight fast of at least 10h, followed by 3 mg BI 409306 PfOS single dose for one day orally with 240 mL of water after an overnight fast of at least 10h.
  Prior to the combined treatment, Fluvoxamine was given for 3 days: 50 mg twice daily on Day -3, followed by 100 mg bid on Day -2 and Day -1.
  There was a washout of at least 6 days after combined administration of BI 409306 and Fluvoxamine in T1.
  Interventions: Drug: Fluvoxamine; Drug: BI 409306 - Powder for oral solution (PfOS)
- 10 mg BI 409306 [R2]/10 mg BI 409306 + 100 mg Fluvoxamine [T2] (Experimental): The subjects were administered 10 mg BI 409306 film-coated tablet single dose for one day in the main phase orally with 240 mL of water after an overnight fast of at least 10h, followed by 10 mg BI 409306 film-coated tablet single dose for one day together with 100 mg Fluvoxamine [Fevarin®] film-coated tablet once daily orally with 240 mL of water after an overnight fast of at least 10h.
  Prior to the combined treatment, Fluvoxamine was given for 3 days: 50 mg twice daily on Day -3, followed by 100 mg bid on Day -2 and Day -1.
  There was a washout of at least 3 days after administration of BI 409306 in R2.
  Interventions: Drug: Fluvoxamine; Drug: BI 409306 - film coated tablet
- 10 mg BI 409306 + 100 mg Fluvoxamine [T2]/10 mg BI 409306 [R2] (Experimental): The subjects were administered 10 mg BI 409306 film-coated tablet single dose for one day in the main phase together with 100 mg Fluvoxamine [Fevarin®] film-coated tablet once daily orally with 240 mL of water after an overnight fast of at least 10h, followed by 10 mg BI 409306 single dose film-coated tablet for one day orally with 240 mL of water after an overnight fast of at least 10h.
  Prior to the combined treatment, Fluvoxamine was given for 3 days: 50 mg twice daily on Day -3, followed by 100 mg bid on Day -2 and Day -1.
  There was a washout of at least 6 days after combined administration of BI 409306 and Fluvoxamine in T2.
  Interventions: Drug: Fluvoxamine; Drug: BI 409306 - film coated tablet

INTERVENTIONS:
Drug: Fluvoxamine — Fluvoxamine
  Other Names: Fevarin®
Drug: BI 409306 - Powder for oral solution (PfOS) — BI 409306 - Powder for oral solution (PfOS)
  Arms: 3 mg BI 409306 + 100 mg Fluvoxamine [T1]/3 mg BI 409306 [R1]; 3 mg BI 409306 [R1]/3 mg BI 409306 + 100 mg Fluvoxamine [T1]
Drug: BI 409306 - film coated tablet — BI 409306 - film coated tablet
  Arms: 10 mg BI 409306 + 100 mg Fluvoxamine [T2]/10 mg BI 409306 [R2]; 10 mg BI 409306 [R2]/10 mg BI 409306 + 100 mg Fluvoxamine [T2]

SUMMARY:
To investigate the influence of fluvoxamine on the pharmacokinetics of BI 409306

ELIGIBILITY:
Inclusion criteria:

* Healthy male or female subjects according to the investigator's assessment, based on a complete medical history including a physical examination, vital signs (BP, PR), 12-lead ECG, and clinical laboratory tests
* Age of 18 to 50 years (incl.)
* BMI of 18.5 to 29.9 kg/m2 (incl.)
* Signed and dated written informed consent prior to admission to the study in accordance with GCP and local legislation
* Male or female subjects who meet any of the following criteria starting from screening until 30 days after trial completion regarding adequate contraception:

  * Non-hormonal intra-uterine device in combination with condom
  * Sexually abstinent
  * Surgically sterilised (including hysterectomy)
  * A vasectomised sexual partner (vasectomy at least 1 year prior to enrolment)
  * Postmenopausal, defined as at least 1 year of spontaneous amenorrhea (in questionable cases a blood sample with simultaneous levels of FSH above 40 U/L and estradiol below 30 ng/L is confirmatory)

Exclusion criteria:

* Any finding in the medical examination (including BP, PR or ECG) is deviating from normal and judged as clinically relevant by the investigator
* Repeated measurement of systolic blood pressure outside the range of 100 to 140 mmHg, diastolic blood pressure outside the range of 60 to 90 mmHg, or pulse rate outside the range of 50 to 85 bpm
* Any laboratory value outside the reference range that the investigator considers to be of clinical relevance
* Any evidence of a concomitant disease judged as clinically relevant by the investigator
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Cholecystectomy and/or surgery of the gastrointestinal tract that could interfere with the pharmacokinetics of the trial medication (except appendectomy and simple hernia repair)
* Diseases of the central nervous system (including but not limited to any kind of seizures or stroke), and other relevant neurological or psychiatric disorders
* History of relevant orthostatic hypotension, fainting spells, or blackouts
* Chronic or relevant acute infections
* History of relevant allergy or hypersensitivity (including allergy to the trial medication or its excipients)
* Use of drugs within 30 days prior to administration of trial medication that might reasonably influence the results of the trial (incl. QT/QTc interval prolongation)
* Participation in another trial where an investigational drug has been administered within 60 days prior to planned administration of trial medication
* Current smoker or ex-smoker who quit smoking less than 30 days prior to screening
* Alcohol abuse (consumption of more than 20 g per day for females and 30 g per day for males)
* Drug abuse or positive drug screening
* Blood donation of more than 100 mL within 30 days prior to administration of trial medication or intended donation during the trial
* Intention to perform excessive physical activities within one week prior to administration of trial medication or during the trial
* Inability to comply with dietary regimen of trial site
* A marked baseline prolongation of QT/QTc interval (such as QTc intervals that are repeatedly greater than 450 ms in males or repeatedly greater than 470 ms in females) or any other relevant ECG finding at screening
* A history of additional risk factors for Torsades de Pointes (such as heart failure, hypokalemia, or family history of Long QT Syndrome)
* Subject is assessed as unsuitable for inclusion by the investigator, for instance, because considered not able to understand and comply with study requirements, or has a condition that would not allow safe participation in the study
* History of major bleeding events (e.g. gastric bleeding, intracranial haemorrhage) based on the investigator's judgement
* Intake of drugs that may interfere with fluvoxamine such as monoamine oxidase inhibitors, and tizanidine.
* Intake of hormonal contraception or ovary hormone replacement therapy in female subjects
* Subjects with a medical history of suicidal behaviour
* History of increased intraocular pressure
* Positive pregnancy test, pregnancy or plans to become pregnant within 30 days after study completion
* Lactation period

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2016-08-25 (Actual); Primary Completion 2016-10-17 (Actual); Study Completion 2016-10-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- Humanpharmakologisches Zentrum Biberach, Biberach, Germany

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization).
  For more details refer to:
  https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- See also: Related Info — http://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This trial was a randomised, open-label, two-treatment, two-sequence, two period crossover trial in healthy male and female subjects in order to compare the test treatment (T1) to the reference treatment (R1) in the pilot phase and the test treatment (T2) to the reference treatment (R2) in the main phase.
  Abbreviations used: R1 (Reference 1), R2 (Reference 2), T1 (Test 1), T2 (Test 2), SD (Standard Deviation).
Groups:
- 3 mg BI 409306 (R1)/3 mg BI 409306 + 100 mg Fluvoxamine (T1): The subjects were administered 3 milligram (mg) BI 409306 Powder for Oral Solution (PfOS) single dose for one day in the pilot phase, taken as 6 mL of 0.5 mg/mL BI 409306 solved in 5 mg/mL (milliliter) tartaric acid orally with 240 mL of water after an overnight fast of at least 10h, followed by 3 mg BI 409306 PfOS single dose for one day together with 100 mg Fluvoxamine (Fevarin®) film-coated tablet once daily orally with 240 mL of water after an overnight fast of at least 10h.
  Prior to the combined treatment, Fluvoxamine was given for 3 days: 50 mg twice daily on Day -3, followed by 100 mg bid on Day -2 and Day -1.
  There was a washout of at least 3 days after administration of BI 409306 in R1.
- 3 mg BI 409306 + 100 mg Fluvoxamine (T1)/3 mg BI 409306 (R1): The subjects were administered 3 mg BI 409306 PfOS single dose for one day in the pilot phase together with 100 mg Fluvoxamine (Fevarin®) film-coated tablet once daily orally with 240 mL of water after an overnight fast of at least 10h, followed by 3 mg BI 409306 PfOS single dose for one day orally with 240 mL of water after an overnight fast of at least 10h.
  Prior to the combined treatment, Fluvoxamine was given for 3 days: 50 mg twice daily on Day -3, followed by 100 mg bid on Day -2 and Day -1.
  There was a washout of at least 6 days after combined administration of BI 409306 and Fluvoxamine in T1.
- 10 mg BI 409306 (R2)/10 mg BI 409306 + 100 mg Fluvoxamine (T2): The subjects were administered 10 mg BI 409306 film-coated tablet single dose for one day in the main phase orally with 240 mL of water after an overnight fast of at least 10h, followed by 10 mg BI 409306 film-coated tablet single dose for one day together with 100 mg Fluvoxamine (Fevarin®) film-coated tablet once daily orally with 240 mL of water after an overnight fast of at least 10h.
  Prior to the combined treatment, Fluvoxamine was given for 3 days: 50 mg twice daily on Day -3, followed by 100 mg bid on Day -2 and Day -1.
  There was a washout of at least 3 days after administration of BI 409306 in R2.
- 10 mg BI 409306 + 100 mg Fluvoxamine (T2)/10 mg BI 409306 (R2): The subjects were administered 10 mg BI 409306 film-coated tablet single dose for one day in the main phase together with 100 mg Fluvoxamine (Fevarin®) film-coated tablet once daily orally with 240 mL of water after an overnight fast of at least 10h, followed by 10 mg BI 409306 single dose film-coated tablet for one day orally with 240 mL of water after an overnight fast of at least 10h.
  Prior to the combined treatment, Fluvoxamine was given for 3 days: 50 mg twice daily on Day -3, followed by 100 mg bid on Day -2 and Day -1.
  There was a washout of at least 6 days after combined administration of BI 409306 and Fluvoxamine in T2.
Period: Period 1
Arm/Group | 3 mg BI 409306 (R1)/3 mg BI 409306 + 100 mg Fluvoxamine (T1) | 3 mg BI 409306 + 100 mg Fluvoxamine (T1)/3 mg BI 409306 (R1) | 10 mg BI 409306 (R2)/10 mg BI 409306 + 100 mg Fluvoxamine (T2) | 10 mg BI 409306 + 100 mg Fluvoxamine (T2)/10 mg BI 409306 (R2)
Started | 2 | 2 | 7 | 7
Completed | 2 | 2 | 7 | 7
Not Completed | 0 | 0 | 0 | 0
Period: Wash-out
Arm/Group | 3 mg BI 409306 (R1)/3 mg BI 409306 + 100 mg Fluvoxamine (T1) | 3 mg BI 409306 + 100 mg Fluvoxamine (T1)/3 mg BI 409306 (R1) | 10 mg BI 409306 (R2)/10 mg BI 409306 + 100 mg Fluvoxamine (T2) | 10 mg BI 409306 + 100 mg Fluvoxamine (T2)/10 mg BI 409306 (R2)
Started | 2 | 2 | 7 | 7
Completed | 2 | 2 | 7 | 6
Not Completed | 0 | 0 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 1
Period: Period 2
Arm/Group | 3 mg BI 409306 (R1)/3 mg BI 409306 + 100 mg Fluvoxamine (T1) | 3 mg BI 409306 + 100 mg Fluvoxamine (T1)/3 mg BI 409306 (R1) | 10 mg BI 409306 (R2)/10 mg BI 409306 + 100 mg Fluvoxamine (T2) | 10 mg BI 409306 + 100 mg Fluvoxamine (T2)/10 mg BI 409306 (R2)
Started | 2 | 2 | 7 | 6
Completed | 2 | 2 | 7 | 6
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Treated Set (TS): This subject set included all subjects in the Randomised Set (all subjects who were randomised, i.e. who had been assigned a study subject number, whether treated or not) who were documented to have received one dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | 3 mg BI 409306 (R1)/3 mg BI 409306 + 100 mg Fluvoxamine (T1) | 3 mg BI 409306 + 100 mg Fluvoxamine (T1)/3 mg BI 409306 (R1) | 10 mg BI 409306 (R2)/10 mg BI 409306 + 100 mg Fluvoxamine (T2) | 10 mg BI 409306 + 100 mg Fluvoxamine (T2)/10 mg BI 409306 (R2) | Total
Number analyzed (Participants) | 2 | 2 | 7 | 7 | 18
Age, Continuous [Mean (Standard Deviation); unit: Years] | 36.0 (5.7) | 41.0 (1.4) | 37.4 (10.6) | 36.9 (6.6) | 37.4 (7.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 2 | 3 | 6
  Male | 2 | 1 | 5 | 4 | 12

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Concentration-time Curve of BI 409306 in Plasma Over the Time Interval From 0 to the Last Quantifiable Data Point (AUC0-tz)
Description: This outcome measured the area under the concentration-time curve of BI 409306 in plasma over the time interval from 0 to the last quantifiable data point (AUC0-tz) in the main phase of the trial (10mg BI 409306 + 100 mg Fluvoxamine (T2) and 10 mg BI 409306 (R2)), as defined in the clinical trial protocol. The statistical model used for the analysis of the endpoint was an ANOVA (Analysis of Variance) model. This model included effects accounting for the following sources of variation: 'sequence', 'subjects within sequences', 'period' and 'treatment'. The effect 'subjects within sequences' was considered as random, whereas the other effects were considered as fixed.
Time Frame: -2:00h (hours: minutes) before drug administration and 0:20h, 0:30h, 0:45h, 1:00h, 1:30h, 2:00h, 2:30h, 3:00h, 4:00h, 6:00h, 8:00h, 10:00h, 12:00h, 24:00h, 34:00h, 48:00h and 72:00h after drug administration.
Population: Pharmacokinetic (PK) analysis set (PKS) restricted to the main phase of the trial: Plasma and urine concentration data and parameters of a subject in the main phase of the trial were included in the statistical PK analyses if they were not flagged for exclusion due to a protocol violation relevant to the evaluation of PK or due to PK non-evaluability.
Measure: Geometric Least Squares Mean (Standard Error); unit: nanomole (nmol)* hour (h)/Liter (L)
Groups:
- 10 mg BI 409306 + 100 mg Fluvoxamine (T2): The subjects were administered 10 mg BI 409306 film-coated tablet single dose for one day together with 100 mg Fluvoxamine (Fevarin®) film-coated tablet once daily orally with 240 mL of water after an overnight fast of at least 10h. Prior to the combined treatment, Fluvoxamine was given for 3 days: 50 mg twice daily on Day -3, followed by 100 mg bid on Day -2 and Day -1.
- 10 mg BI 409306 (R2): The subjects were administered 10 mg BI 409306 film-coated tablet single dose for one day orally with 240 mL of water after an overnight fast of at least 10h.
Arm/Group | 10 mg BI 409306 + 100 mg Fluvoxamine (T2) | 10 mg BI 409306 (R2)
Number analyzed (Participants) | 14 | 13
nanomole (nmol)* hour (h)/Liter (L) | 5441.83 (NA) — Adjusted geometric standard error = 1.178 | 175.10 (NA) — Adjusted geometric standard error = 1.184
Statistical Analysis 1: Comparison: 10 mg BI 409306 + 100 mg Fluvoxamine (T2) vs 10 mg BI 409306 (R2); The statistical model used for the analysis of the endpoint was an ANOVA (Analysis of Variance) model. This model included effects accounting for the following sources of variation: 'sequence', 'subjects within sequences', 'period' and 'treatment'. The effect 'subjects within sequences' was considered as random, whereas the other effects were considered as fixed; Test type: Other; Adjusted geometric Mean ratio [%] = 3107.80, 90% CI 2-sided [2332.90 to 4140.10] — The estimated parameter was the adjusted geometric Mean (gMean) ratio [%] = adjusted gMean T2/ adjusted gMean R2. Intra-individual geometric coefficient of variation [%] =42.7

2. Primary Outcome: Maximum Measured Concentration of BI 409306 in Plasma (Cmax)
Description: This outcome measure presents the maximum measured concentration of BI 409306 in plasma in the main phase of the trial (10mg BI 409306 + 100 mg Fluvoxamine (T2) and 10 mg BI 409306 (R2)), as defined in the clinical trial protocol. The statistical model used for the analysis of the endpoint was an ANOVA (Analysis of Variance) model. This model included effects accounting for the following sources of variation: 'sequence', 'subjects within sequences', 'period' and 'treatment'. The effect 'subjects within sequences' was considered as random, whereas the other effects were considered as fixed.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Least Squares Mean (Standard Error); unit: nmol/L
Arm/Group | 10 mg BI 409306 + 100 mg Fluvoxamine (T2) | 10 mg BI 409306 (R2)
Number analyzed (Participants) | 14 | 13
nmol/L | 660.011 (NA) — Adjusted geometric standard error = 1.136 | 100.153 (NA) — Adjusted geometric standard error = 1.143
Statistical Analysis 1: Comparison: 10 mg BI 409306 + 100 mg Fluvoxamine (T2) vs 10 mg BI 409306 (R2); [analysis description as in outcome 1, analysis 1]; Test type: Other; Adjusted geometric Mean ratio [%] = 659.00, 90% CI 2-sided [489.791 to 886.676] — The estimated parameter was the adjusted geometric Mean (gMean) ratio [%] = adjusted gMean T2/ adjusted gMean R2. Intra-individual geometric coefficient of variation [%]=44.8

3. Secondary Outcome: Area Under the Concentration-time Curve of BI 409306 in Plasma Over the Time Interval From 0 Extrapolated to Infinity (AUC 0-infinity)
Description: This outcome measure presents AUC0-infinity (area under the concentration-time curve of BI 409306 in plasma over the time interval from 0 extrapolated to infinity) in the main phase of the trial (10mg BI 409306 + 100 mg Fluvoxamine (T2) and 10 mg BI 409306 (R2)), as defined in the clinical trial protocol. The statistical model used for the analysis of the endpoint was an ANOVA (Analysis of Variance) model. This model included effects accounting for the following sources of variation: 'sequence', 'subjects within sequences', 'period' and 'treatment'. The effect 'subjects within sequences' was considered as random, whereas the other effects were considered as fixed.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Least Squares Mean (Standard Error); unit: nmol*h/L
Arm/Group | 10 mg BI 409306 + 100 mg Fluvoxamine (T2) | 10 mg BI 409306 (R2)
Number analyzed (Participants) | 14 | 13
nmol*h/L | 5450.03 (NA) — Adjusted geometric standard error = 1.178 | 175.61 (NA) — Adjusted geometric standard error = 1.184
Statistical Analysis 1: Comparison: 10 mg BI 409306 + 100 mg Fluvoxamine (T2) vs 10 mg BI 409306 (R2); [analysis description as in outcome 1, analysis 1]; Test type: Other; Adjusted geometric Mean ratio [%] = 3103.41, 90% CI 2-sided [2330.50 to 4132.65] — [estimate comment as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: From first drug administration until 4 days after last drug, up to 8.71 weeks.
Description: Treated Set (TS): This subject set included all subjects in the Randomised Set (all subjects who were randomised, i.e. who had been assigned a study subject number, whether treated or not) who were documented to have received one dose of study drug.
Groups:
- 3 mg BI 409306 (R1): The subjects were administered 3 mg BI 409306 PfOS orally with 240 mL of water after an overnight fast of at least 10h. The Adverse Event (AE) assignment period for this treatment lasted from the time of the administration of the single dose of BI 409306 until the end of the Residual Effect Period (REP) (24h).
- Pilot Phase: Loading Fluvoxamine: The subjects were administered Fluvoxamine over 3 days orally with 240 mL of water after an overnight fast of at least 10h. The AE assignment period for this treatment lasted from the first Fluvoxamine dose given over 3 days and ended with the time of the administration of a single dose of BI 409306 together with Fluvoxamine.
- 3 mg BI 409306 + 100 mg Fluvoxamine (T1): The subjects were administered 3 mg BI 409306 PfOS single dose for one day together with 100 mg Fluvoxamine (Fevarin®) film-coated tablet orally with 240 mL of water after an overnight fast of at least 10h. The AE assignment period for this treatment lasted from the time of the administration of the single dose of BI 409306 together with Fluvoxamine till the end of the REP (96h).
- 10 mg BI 409306 (R2): The subjects were administered 10 mg BI 409306 film-coated tablet single dose orally with 240 mL of water after an overnight fast of at least 10h for one day. The AE assignment period for this treatment lasted from the time of the administration of the single dose of BI 409306 until the end of the REP (24h).
- Main Phase: Loading Fluvoxamine: The subjects were administered Fluvoxamine over 3 days orally with 240 mL of water after an overnight fast of at least 10h. The AE assignment period for this treatment lasted from the time of the administration of the Fluvoxamine dose given over 3 days and ended with the time of the administration of a single dose of BI 409306 together with Fluvoxamine.
- 10 mg BI 409306 + 100 mg Fluvoxamine (T2): The subjects were administered 10 mg BI 409306 film-coated tablet single dose for one day together with 100 mg Fluvoxamine (Fevarin®) film-coated tablet orally with 240 mL of water after an overnight fast of at least 10h. The AE assignment period for this treatment lasted from the time of the administration of a single dose of BI 409306 together with Fluvoxamine till the end of the REP (96h).
Arm/Group | 3 mg BI 409306 (R1) | Pilot Phase: Loading Fluvoxamine | 3 mg BI 409306 + 100 mg Fluvoxamine (T1) | 10 mg BI 409306 (R2) | Main Phase: Loading Fluvoxamine | 10 mg BI 409306 + 100 mg Fluvoxamine (T2)
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/4 | 0/4 | 0/13 | 0/14 | 0/14
Other Adverse Events (participants affected / at risk) | 0/4 | 3/4 | 1/4 | 0/13 | 10/14 | 3/14
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 3 mg BI 409306 (R1) (N=4) | Pilot Phase: Loading Fluvoxamine (N=4) | 3 mg BI 409306 + 100 mg Fluvoxamine (T1) (N=4) | 10 mg BI 409306 (R2) (N=13) | Main Phase: Loading Fluvoxamine (N=14) | 10 mg BI 409306 + 100 mg Fluvoxamine (T2) (N=14)
Dry eye (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0
Aphthous ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Hypoaesthesia oral (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 4 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Sluggishness (General disorders) | 0 | 1 | 0 | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 0 | 0 | 2 | 0
Headache (Nervous system disorders) | 0 | 1 | 0 | 0 | 3 | 1
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes